CLINICAL TRIAL: NCT06610721
Title: 'Improving Urinary Tract Infection Diagnosis in Older Patients: Validation of a Biomarker Panel (UTI-GOLD)'
Acronym: UTI-GOLD
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Nora El Moussaoui, drs. N. El Moussaoui, Leiden University Medical Center
Other Study IDs: nWMODIV2_2024025
Record Dates: First submitted 2024-09-19; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Urinary Tract Infection (Diagnosis)
Keywords: Urinary tract infection; Biomarkers
MeSH Terms: conditions — Urinary Tract Infections; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly patients with a suspected urinary tract infection
  Interventions: Diagnostic Test: Urine Biomarkers

INTERVENTIONS:
Diagnostic Test: Urine Biomarkers — At baseline midstream urine will be collected in a sterile urine container.

SUMMARY:
The goal of this study is to improve the diagnosis of urinary tract infections (UTI) in older people (≥65 years). The main research questions are:

Research questions

* What is the optimal cut-off for each individual biomarker NGAL,IL-6,AZU,TIMP2 and CXCL9 and associated, sensitivity, specificity, negative and positive predictive value.
* sensitivity, specificity, negative and positive predictive value of a urine leukocyte count cut-off of 200 cells/microL (validation)
* What is the optimal combination of biomarkers for UTI diagnosis in older patients
* As a secondary objective this study aims to evaluate the association between the levels of individual biomarker levels and 1) duration of symptoms 2) complications, 3) recurrence of UTI within 2 months, and length of hospital stay. Next to this, the performance of the astrego PA100 will be validated in diagnosing bacteriuria.

Participants will:

* be asked to provide a urine sample once at the beginning of the study
* be asked to answer some questions about their symptoms and overall health at the beginning of the study and after 8 weeks
* have their vital parameters (temperature and blood pressure) measured once at the beginning of the study

ELIGIBILITY:
Inclusion criteria:

* Age 65 years or older
* Clinically suspected UTI by treating physician
* Sufficient understanding of the Dutch language

Exclusion criteria:

* Inability to obtain urine
* Inability to provide written consent
* The presence of an indwelling catheter

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be recruited in the hospital setting, long term care and general practice. Patients will be recruited through an existing network of hospitals, primary care offices and long stay facilities in the Leiden and the Hague region (the Netherlands). Additionally, there is a collaboration with university college hospital in London (the UK).
  Patients with suspected UTI in these centers will be identified by their attending healthcare provider. The attending healthcare provider will notify the study team, who will proceed the inclusion process.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of individual urine biomarkers | At Baseline
  Sensitivity and specificity in percentages for the different biomarkers include; NGAL, IL-6, AZU, TIMP2 and CXCL9.
Diagnostic accuracy of individual urine biomarkers | At Baseline
  Positive and negative predictive value in percentages for the different biomarkers include; NGAL, IL-6, AZU, TIMP2 and CXCL9.
Diagnostic accuracy of individual urine biomarkers | At Baseline
  Likelihood ratios for the different biomarkers include; NGAL, IL-6, AZU, TIMP2 and CXCL9.
Diagnostic accuracy of individual urine biomarkers | At Baseline
  Area under the receiver operating characteristic curve (AUC) for the different biomarkers include; NGAL, IL-6, AZU, TIMP2 and CXCL9.
Diagnostic accuracy of urine biomarker panel | At Baseline
  Sensitivity and specificity in percentages for the optimal combination of biomarkers
Diagnostic accuracy of urine biomarker panel | At Baseline
  positive and negative predictive values in percentages for the optimal combination of biomarkers.
Diagnostic accuracy of urine biomarker panel | At Baseline
  The likelihood ratios for the optimal combination of biomarkers.
Diagnostic accuracy of urine biomarker panel | At Baseline
  The area under the receiver operating characteristic curve (AUC) for the optimal combination of biomarkers.
Diagnostic accuracy of leukocytes in urine | At Baseline
  Sensitivity and specificity in percentages for the cut-off of 200 leukocytes/microL in urine.
Diagnostic accuracy of leukocytes in urine | At Baseline
  Negative and positive predictive value in percentages for the cut-off of 200 leukocytes/microL in urine

SECONDARY OUTCOMES:
Duration of symptoms | 1 week after inclusion, if not yet resolved again at 8 weeks
Length of hospital stay | 1 week after inclusion, if not yet resolved again at 8 weeks
Complications | 1 week after inclusion, if not yet resolved again at 8 weeks
Recurrence of UTI <2 months | 8 weeks after inclusion
Diagnostic performance of PA100 in detecting bacteruria | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden university medical center (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
data will be shared in a registry. after completion of the study. The data sharing plan will be developed
Supporting Information: Study Protocol
Time Frame: to be determined
Access Criteria: to be determined

REFERENCES:
- [Derived] El Moussaoui N, van Andel E, van der Beek MT, Vlot JA, Bilsen MP, van Nieuwkoop C, Lauw FN, Delfos NM, Stalenhoef JE, Sijbom M, Akintola AA, Achterberg WP, Goeman JJ, Leyten EMS, van Uhm JIM, Corstjens PLAM, Mooijaart SP, Conroy SP, Cobbaert CM, Visser LG, Lambregts MMC. Validation of urinary biomarkers for accurate diagnosis of urinary tract infections in older adults across primary care, hospitals and long-term care facilities in the Netherlands and UK (UTI-GOLD): a multicentre observational study protocol. BMJ Open. 2025 Jun 18;15(6):e103311. doi: 10.1136/bmjopen-2025-103311. PMID 40533212